CLINICAL TRIAL: NCT05295667
Title: Combination of Doppler Measurements With Amniotic Fluid Volume for the Predicition of Perinatal Outcome in FGR
Brief Title: Doppler and AFV for Outcome Prediction ın FGR
Status: Completed | Type: Observational
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, Associated Proffesor, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Other Study IDs: Besimoglu01
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fetal Growth Retardation Group
  Interventions: Diagnostic Test: Doppler measurement in combination with amniotic fluid volume

INTERVENTIONS:
Diagnostic Test: Doppler measurement in combination with amniotic fluid volume — Ultrasonographic evaluation

SUMMARY:
The investigator contrived a prospective study of AUCR to compare its association to adverse perinatal outcomes with other established doppler parameters, such as CPR and UCR within a population of suspected FGR fetuses at term.

ELIGIBILITY:
Inclusion Criteria:

* SİNGLETON PREGNANCİES WİTH FGR FETUSES
* AFTER 37th GESTATİONAL WEEKS

Exclusion Criteria:

* SİNGLE OR MUTİPL FETAL ANOMALİES
* EVİDENCE OF İNTRAUTERİNE ENFECTİON

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant women with fetal growth retardation (FGR)
Study Population: A pregnant womens between 18-40 years of age with singleton pregnancy after 37 weeks of gestational age with FGR
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
the prediction power of adverse perinatal outcome with new doppler parameters ( such as AUCR) | 1 year
  enterence to neonatal intensive care unit and severe fetal acidemia ( pH: >7.10)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stumpfe FM, Faschingbauer F, Kehl S, Pretscher J, Emons J, Gass P, Mayr A, Schmid M, Beckmann MW, Stelzl P. Amniotic-Umbilical-to-Cerebral Ratio - A Novel Ratio Combining Doppler Parameters and Amniotic Fluid Volume to Predict Adverse Perinatal Outcome in SGA Fetuses At Term. Ultraschall Med. 2022 Apr;43(2):159-167. doi: 10.1055/a-1205-0161. Epub 2020 Jul 28. PMID 32722822